CLINICAL TRIAL: NCT03089580
Title: Intense Pulsed Light Study for Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eversight Michigan/Michigan Eye Bank (Unknown)
Responsible Party: Principal Investigator, Sarah Wood, Ophthalmology, Instructor in Ophthalmology and Visual Sciences, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00119518
Record Dates: First submitted 2017-03-13; First posted 2017-03-24 (Actual); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Dry Eyes Chronic
MeSH Terms: interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intense Pulsed Light Treatment (Experimental): Participants will have one eye randomized to receive the intense pulsed light (IPL) therapy treatment while their other eye will receive the sham treatment. Participants will receive approximately 15 light spots to areas around the eye, lower eyelid, cheek, side of the nose and temple. The energy level will be based on skin type. IPL will be administered 4 times throughout the study.
  Interventions: Device: Intense Pulsed Light Therapy
- Sham Treatment (Placebo Comparator): Participants will have the other eye randomized to receive a sham treatment. The sham treatment will be conducted by placing the intense pulsed light (IPL) device to approximately 15 areas around the eye, lower eyelid, cheek, side of nose and temple without delivery of the light. The sham treatment will mimic the IPL treatment but no light will be delivered. Sham treatment will be administered 4 times throughout the study.
  Interventions: Procedure: Sham Treatment

INTERVENTIONS:
Device: Intense Pulsed Light Therapy — Intense pulsed light therapy is a non-invasive and non-laser light treatment that was approved in 1995 by the FDA for dermatology. Participants will receive a total of 4 treatments over the course of the study.
  Arms: Intense Pulsed Light Treatment
Procedure: Sham Treatment — The sham treatment will mimic the IPL treatment but no light will be delivered. Sham treatment will be administered 4 times throughout the study.
  Arms: Sham Treatment

SUMMARY:
This study will evaluate the efficacy of intense pulsed light (IPL) therapy for the treatment of dry eye disease. One eye of the participant will be randomized to receive the IPL treatment.

DETAILED DESCRIPTION:
Dry eye disease (DED) affects tears and the front surface of the eye. Patients who have DED can experience symptoms of discomfort, blurry vision, redness, and pain. DED can also cause tears to become unstable which could result in damage to the front surface of the eye.

There are two types of DED. The one the investigators are studying is called evaporative dry eye disease. This type of DED occurs because the pores on the eyelids are not functioning properly. In preliminary studies, a new treatment called Intense Pulsed Light (IPL) has shown promise to reduce signs and symptoms of evaporative DED. IPL is a non-invasive and non-laser light treatment that was approved in 1995 by the FDA for dermatology. It is commonly used for treatment of facial rosacea, acne, and hair, wrinkle and lesion removal. It is not currently approved for the treatment of dry eye disease. This treatment is thought to provide relief of evaporative DED symptoms and improve the expression of the pores on the edge of the eyelid.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent;
* Diagnosed with evaporative dry eye disease with symptoms for 6 months or more;
* Able and willing to comply with follow-up visits, phone calls and intense pulsed light treatments;
* Agree to using an effective method of birth control during the course of the study;
* Agree to continue current dry eye treatments during the course of the study;
* Fitzpatrick skin scale of 1 (very fair) to 4 (olive) as determined by an investigator.

Exclusion Criteria:

* Darker skinned individuals defined by the Fitzpatrick scale 5 and 6 as determined by an investigator;
* Neurotrophic keratitis;
* Ectropion, trauma, or any other lid abnormalities;
* Previous diagnosis of Stevens Johnson syndrome or graft versus host disease;
* Ocular burn, active ocular infection, or active ocular inflammation;
* Currently pregnant or trying to become pregnant in the next 5 months;
* Systemic conditions or currently taking medications which makes light therapy contraindicated (the use of doxycycline is allowed);
* Tattoos in the treatment area;
* Patients who have had intense pulsed light therapy, Lipiflow or Meibothermoflo within the past six months;
* Contact lens wear more than one time/week or history of refractive surgery;
* Glaucoma drop use
* Ophthalmic steroid use within the past 30 days;
* Punctal plugs if instilled within 30 days of the start of the study;
* Obvious asymmetry between the two eyes deemed significant by the investigators (such as punctal plugs or cautery in only one eye, etc);
* History of a trabeculectomy or tube surgery;
* Uncontrolled ocular or systemic disease;
* Ocular or eyelid surgery within the last 6 months;
* Any condition which leads the investigator to believe that the patient cannot comply with the study requirements and/or the patient may be placed at risk with participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-03-25 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Wood, OD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Kellogg Eye Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 participants were recruited. Each participant received the Intense Pulse Light treatment in one eye and the sham treatment in their other eye.
Units Other Than Participants: Eyes
Groups:
- Intense Pulsed Light Treatment: Participants had one eye randomized to receive the intense pulsed light (IPL) therapy treatment in the right or left eye, while their other eye received the sham treatment. 14 eyes received IPL, and 14 eyes received the sham treatment. Throughout the study, the IPL treatment eye was always the same for each individual.
  Participants received approximately 15 light spots to areas around the eye, lower eyelid, cheek, side of the nose and temple. The energy level was based on skin type. IPL was administered 4 times throughout the study.
  Intense Pulsed Light Therapy: Intense pulsed light therapy is a non-invasive and non-laser light treatment that was approved in 1995 by the FDA for dermatology. Participants received a total of 4 treatments over the course of the study.
Period: Overall Study
Arm/Group | Intense Pulsed Light Treatment
Started | 14; 28 Eyes
Completed | 12; 24 Eyes
Not Completed | 2; 4 Eyes
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intense Pulsed Light Treatment
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Tear Breakup Time Average
Description: Three tear breakup time measurements will be taken of each eye. The averages of those eyes treated with intense pulsed light treatment will be compared to those eyes that received the sham treatment.
Time Frame: 16.5 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Sham Treatment: Participants had one eye randomized to receive the intense pulsed light (IPL) therapy treatment in the right or left eye, while their other eye received the sham treatment. 14 eyes received IPL, and 14 eyes received the sham treatment. Throughout the study, the IPL treatment eye was always the same for each individual.
  Participants received approximately 15 light spots to areas around the eye, lower eyelid, cheek, side of the nose and temple. The energy level was based on skin type. IPL was administered 4 times throughout the study.
  Intense Pulsed Light Therapy: Intense pulsed light therapy is a non-invasive and non-laser light treatment that was approved in 1995 by the FDA for dermatology. Participants received a total of 4 treatments over the course of the study.
Arm/Group | Intense Pulsed Light Treatment | Sham Treatment
Number analyzed (Participants) | 14 | 14
Seconds
  Visit 1 at Baseline | 3.3 (1.3) | 3.0 (1.5)
  Visit 5 at 16.5 Weeks | 4.1 (2.3) | 4.5 (2.5)
Statistical Analysis 1: Comparison: Intense Pulsed Light Treatment vs Sham Treatment; The primary study outcome of pre to post change in TBUT within the treated eye and also the untreated, control eye dictated the use of a paired statistical approach to sample size estimation. Clinically relevant pre to post TBUT increase of 3 seconds with a standard deviation of 4.5 seconds was used. Type I and II error estimates used were standard for a non-pivotal study, 0.05 & 0.20. The estimated the sample size needed detect this difference in TBUT is 27 subjects; Test type: Superiority — Paired, Student's t-test was used to contrast the outcome variable of TBUT in the treated eye versus the sham eye from visit 1 to visit 5. The null hypothesis to be tested is one of no change from pre- to post treatment, with a Type I error probability of 0.05 for the primary outcome assessment. The pattern of change over the 4 treatment visits in these continuous variables will be assessed using mixed, linear regression. SAS version 9.4 statistical software (SAS Institute, Cary, NC) was used; p = 0.3, paired t test

2. Primary Outcome: Change in Scores of the Ocular Surface Disease Index Questionnaire
Description: Patients completed the Ocular Surface Disease Index Questionnaire at each visit before they received the IPL and sham treatments. The questionnaire is assessed on a scale of 0 to 100 with 0 meaning normal and the higher scores representing greater dry eye disease severity. This questionnaire has been validated to assess ocular symptoms for a patient but cannot be separated by eye. Therefore, the results cannot be given by treatment vs. sham, but for the participant overall.
Time Frame: 7 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intense Pulsed Light Treatment
Number analyzed (Participants) | 14
score on a scale
  Visit 1 at Baseline | 29.7 (21.6)
  Visit 2 at 4 weeks | 25.6 (17.2)
  Visit 3 at 8 weeks | 23.6 (20.1)
  Visit 4 at 12 weeks | 20.7 (18.6)
  Visit 5 at 16.5 weeks | 23.7 (19.8)
  7 month phone call | 22.2 (19.5)
Statistical Analysis 1: Comparison: Intense Pulsed Light Treatment; Test type: Superiority — The p-value results from a test of the hypothesis that the change in OSDI from visit 1 does not differ from zero. Change distributions that met normal distribution test criteria (Shapiro-Wilk p-value >0.05) were tested with the paired Student's t-test; non-normal change distributions (at visits 2 & 4) were tested with the non-parametric Wilcoxon signed rank test; p = 0.2026, paired t test

ADVERSE EVENTS:
Time Frame: 7 months
Description: Adverse events for either eye were determined by the investigator as "possibly", "probably" or "definitely" related to the IPL treatment or study procedures
Groups:
- Intense Pulsed Light Treatment: Participants will have one eye randomized to receive the intense pulsed light (IPL) therapy treatment and will receive the sham treatment in their other eye.
  Participants will receive approximately 15 light spots to areas around the eye, lower eyelid, cheek, side of the nose and temple. The energy level will be based on skin type. IPL will be administered 4 times throughout the study.
  Intense Pulsed Light Therapy: Intense pulsed light therapy is a non-invasive and non-laser light treatment that was approved in 1995 by the FDA for dermatology. Participants will receive a total of 4 treatments over the course of the study.
Arm/Group | Intense Pulsed Light Treatment | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intense Pulsed Light Treatment (N=14) | Sham Treatment (N=14)
Subconjunctival Hemorrhage (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT03089580/Prot_SAP_000.pdf